CLINICAL TRIAL: NCT06945679
Title: Effects of Carica Papaya Leaf Extract (CPLE) in the Outcome of Hospitalized Dengue Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Institute of Technology Transfer & Innovation (ITTI) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Shohael Mahmud Arafat, Professor, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSMMU/2024/3129
Record Dates: First submitted 2025-03-22; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPLE group (Active Comparator): After confirming the diagnosis of Dengue fever,the potential benefits and risks of the use of CPLE in capsule form will be explained to the patients.Patients will be properly explained about purpose and procedure of the study.After taking informed written consent, 168 patients with dengue fever will be finally enrolled in the study.Then total 168 patients will be randomized into 2 groups by using website www.randomization.com. It will be a double-blind study,CPLE and Placebo will be marked as either Group A or Group B.Half of the patients will receive Group A and other half will receive Group B drug along with standard treatment according to national guideline,Each participant will receive either CPLE or Placebo,500 mg 2 capsules three times daily for 5 days and will be followed up daily upto study day 5.
  Interventions: Drug: CPLE
- Placebo (Placebo Comparator): he patients will be assigned to one of the two treatment arms:
  1. Active drug: CPLE 500mg 2 capsule t.i.d for 5 days
  2. Placebo: visually matched placebo 2 capsule t.i.d for 5 days The oral capsule of CPLE and placebo will be provided by the Institute of Technology Transfer and Innovation (ITTI), an institute in Bangladesh Council of Scientific and Industrial Research (BCSIR). On receipt, the medications will be stored in a secure area at room temperature. Enrolled patients will receive CPLE or placebo for 5 days.
  Clinical data will be captured on structured case report forms.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPLE — It will be a double-blind study,CPLE and Placebo will be marked as either Group A or Group B.Half of the patients will receive Group A and other half will receive Group B drug along with standard treatment according to national guideline,Each participant will receive either CPLE or Placebo,500 mg 2 capsules three times daily for 5 days and will be followed up daily upto study day 5.
  Arms: CPLE group
Drug: Placebo — The patients will be assigned to visually matched placebo 2 capsule t.i.d for 5 days The oral capsule of CPLE and placebo will be provided by the Institute of Technology Transfer and Innovation (ITTI), an institute in Bangladesh Council of Scientific and Industrial Research (BCSIR). On receipt, the medications will be stored in a secure area at room temperature. Enrolled patients will receive CPLE or placebo for 5 days.
  Clinical data will be captured on structured case report forms.
  Arms: Placebo

SUMMARY:
Its a double-blind placebo controlled multicenter study involving confirmed dengue patients who are hospitalized.168 Patients will be enrolled according to specific inclusion & exclusion criteria and they will be divided into two equal arms..After taking informed written consent patients will be provided with either CPLE 500 mg 2 capsule 3 times daily for 5 days or placebo and they will be followed up upto discharge from hospital or ICU transfer or death.

We want to see the effects of CPLE in the outcome of hospitalized dengue patients in comparison to placebo group.

Participants will be asked to take oral CPLE or placebo 500 mg 2 capsules 3 times daily for 5 days.

DETAILED DESCRIPTION:
Dengue, an important viral diseases of human, has become a life-threatening condition in recent decades. It is found in tropical and subtropical regions worldwide, mostly in urban area. Dengue, a Flaviviridae virus, is transmitted through Aedes agypti mosquito. 5-7 days after an infected mosquito bites, a healthy person may be affected by Dengue. Usual symptoms of Dengue fever include high fever, rash, and headaches as well as muscle and joint pain, eye pain, vomiting, and nausea, diarrhoea. It has four serotypes (Dengue virus-1 to Dengue virus-4) and an individual can be infected multiple times due to the different virus types which can result in a severe form of dengue known as dengue hemorrhagic fever (DHF). It has been estimated that there are about 50-100 million cases of dengue fever (DF) and 500,000 cases of dengue hemorrhagic fever (DHF) every year. Thrombocytopenia is very common in dengue fever. Thrombocytopenia in dengue may be developed by the down regulation of platelet production in bone marrow, the destruction of existing platelets, the production of antibodies against platelets and the clearance of platelets mediated by these antibodies. There is no specific treatment for dengue; only supportive care is given for management. Hypotension, thrombocytopenia, and hemoconcentration during the febrile phase might indicate progression towards severe disease. The thrombocytopenia can lead to mortality if left unattended or untreated.Till now there is no approved vaccine or drug against dengue virus, therefore there is an urgent need of development of alternative solutions for dengue. Several plants species have anti-dengue activity. Traditional medicinal plants have antiviral activity and some are used to treat viral infections in animals and humans.Carica papaya has significant platelet augmentation activity. So Carica Papaya leaf extract can be used as supportive treatment for thrombocytopenic disorders and dengue hemorrhagic fever which may be an alternative to platelet transfusions. The prevalence and incidence of dengue fever and death due to its complications have been increased drastically in these recent years in Bangladesh. Till now there is no established specific and effective treatment by synthetic medicines. But, Malaysia effectively controlled its incidences and death of patients using Carica papaya leaves along with proper supportive care and hospitalization.There are several studies regarding usefulness of herbal medicine in Dengue fever. Researchers found that Carica papaya leaf extract helps to increase the platelet count and also have beneficial effects in these patients.It is effective and safe for the dengue patients.Carica papaya leaf extract has antiviral activities, can prevent thrombocytopenia and can improve the immunity during dengue fever. It can acts as a strong stimulant of IL-6 and SCF (Stem Cell Factor) might help to raise the platelet counts in infected patients. CPLE, rich in papain, which also raises thrombocyte (platelet) count in dengue patients. The qualitative phytochemical analysis reveals that except steroids and tannins all the phytochemical including glycosides, alkaloids, saponins, flavonoids, proteins are present in leaf of papaya. Papaya leaf contains anti-oxidant vitamins and minerals which may help to increase the hemoglobin,hematocrit, Red blood cells, thrombocytes and total protein contents. CPLE prevents stress-induced destruction of the plasma membrane. Flavonoids and other phenolic compounds present in papaya leaf extracts were responsible for membrane stabilizing property and thereby prevent the internal bleeding. A recent study showed that flavonoids, present in Carica papaya inhibits NS2B-NS3 protease which can prevent the DEN-2 Virus assembly.

Till now there is no specific treatment of Dengue virus infection while there is no effective antiviral drug, only symptomatic and supportive care is given as the main forms of treatment. Dengue induced thrombocytopenia is the most important complication of dengue,so prevention of thrombocytopenia and increasing the platelet count may improve the outcome of the dengue patients.Eltrombopeg and corticosteroids are effectively used in some diseases to increase the platelet count.Eltrombopeg is an expensive drug and its' use in dengue fever is not established yet.Use of corticosteroid in dengue fever is under trial. Sometimes platelet transfusion is needed to prevent thrombocytopenia induced complications and reduce dengue related mortality. But processing of platelet transfusion is expensive and platelet transfusion machine is not available at distant places in our country. So it is not possible to transfuse platelet to the patients with thrombocytopenia at distant places .Many studies on herbal medicine have suggested that Carica Papaya has a potential role in increasing platelet count by increasing megakaryopoiesis, decreasing platelet destruction by membrane stabilization, decreasing viral assembly and platelet aggregation. It has been demonstrated that CPLE increases platelet counts in patients with thrombocytopenia safely and effectively though some studies gave controversial report. Moreover,it has not yet been determined how effective CPLE is at reducing the severity of dengue fever.Some countries like Malaysia is already using CPLE effectively in dengue patients.But data regarding this condition is very scarce.I want to see whether the CPLE effectively improves the outcome of dengue patients by increasing platelet counts,lowering the requirement for platelet transfusions,reducing the bleeding episodes,hospital stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are confirmed dengue fever by positive NS1 dengue Antigen and/ Dengue IgM antibody.
2. Day of illness ≤ 5 days

Exclusion Criteria:

1. Children (<18 years)
2. Patients already getting Papaya
3. Currently pregnant or lactating
4. Patients on steroids or any immunosuppressant
5. Patients who received platelet transfusion during the same admission
6. Patient with known causes of thrombocytopenia
7. Patients with alanine aminotransferase (ALT) levels >150 U/L
8. Patient with serum creatinine >1.4 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Rise in platelet count | 5 days
  The treatment and placebo groups will compare the peak platelet count

SECONDARY OUTCOMES:
Return of hematocrit levels towards baseline | 5 days
  The treatment and placebo groups will compare the normalization of hematocrit value

OTHER OUTCOMES:
Bleeding Manifestations | six days
  The frequency of bleeding events determined by clinical evaluation between the treatment and placebo groups

CONTACTS AND LOCATIONS:
Locations (1):
- Prof Shohael Mahmud Arafat, Dhaka, Dhaka Division, Bangladesh